CLINICAL TRIAL: NCT04592497
Title: Evaluation of the Safety and Performance of the Very High Power-Short Duration QDOT Strategy in Patients Referred for Atrial Fibrillation Ablation.
Brief Title: Evaluation of the Safety and Performance of the Very High Power-Short Duration QDOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, PI, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-20-EC-488
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QDOT (Experimental): will undergo the AF ablation procedure with assistance THERMOCOOL SMARTTOUCH SF-5D QDOT system
  Interventions: Procedure: AF ablation
- standard (Active Comparator): will undergo the AF ablation procedure with assistance standard Thermocool Smartouch SF system
  Interventions: Procedure: AF ablation

INTERVENTIONS:
Procedure: AF ablation — Prospective, single-center, non-randomized, open label, two arm study. After informed consent, 60 consecutive subjects who are scheduled to undergo AF ablation will be enrolled in the study in two equally sized groups of 30 subjects each. One group will undergo the procedure with assistance THERMOCOOL SMARTTOUCH SF-5D QDOT system and the other with the standard Thermocool Smartouch SF system. Data will be collected from all subjects during the ablation procedure and post procedure for a period of 12 months. Data will be anonymized by removing patient protected health information, only initials will be used.

SUMMARY:
The aim of the present study is to compare the safety and short-term performance between THERMOCOOL SMARTTOUCH SF-5D QDOT system used with fast ablation mode and the standard Thermocool Smartouch SF in treatment of patients with atrial fibrillation (AF).

DETAILED DESCRIPTION:
The very high power-short duration (vHPSD) catheter, is a novel CF catheter optimized for temperature-controlled ablation with microelectrodes and 6 thermocouples for real-time temperature monitoring during ablation. The associated vHPSD algorithm modulates power to maintain target temperature during these vHPSD lesions (90 W, 4 s). In preclinical models, vHPSD ablation with this novel catheter has improved atrial linear lesion contiguity, transmurality, and durability and has substantially reduced radiofrequency ablation times, but with a safety profile similar to those of standard irrigated radiofrequency ablation catheters.

The QDOT -FAST study demonstrated the clinical feasibility and safety of vHPSD ablation. Procedure and fluoroscopy times were substantially lower than historical standard ablation with point-by-point catheters.

The aim of the present study is to compare the safety and short-term performance between THERMOCOOL SMARTTOUCH SF-5D QDOT system used with fast ablation mode and the standard Thermocool Smartouch SF in treatment of patients with atrial fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

* Male and female >18 years old.
* Subjects must provide written informed consent to participate in the study.
* Subject is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations.

Exclusion Criteria:

* Pregnant women.
* Patients with iodine contrast media allergy
* Patients with renal failure (GFR <60ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
procedure time | 1 day
  The procedural and fluoroscopy time required for the procedure (in minutes).
isolation efficacy | 1 day
  The first time pulmonary vein isolation (percentages of success)
Recurrence of AF | 1 year
  Recurrence of AF (will be assessed by Holter monitoring)

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Chorin, MD PhD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
The results of the study will be submitted to a peer-reviewed journal in the field of cardiac arrhythmia